CLINICAL TRIAL: NCT01938469
Title: Effect of Meal Number, Frequency, and Form on Satiety and Metabolism After Weight Loss Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-117
Record Dates: First submitted 2013-08-21; First posted 2013-09-10 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Gastric Bypass Surgery; Obesity
Keywords: Bariatric; Gastric Bypass; Gastric Banding,; Incretins; glucagon-like peptide-1(GLP-1); gastric inhibitory peptide (GIP)
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solid Meal (Other): Participants in this group will be administered only solid meals on both study visits completed before surgery (T0) and 12-15 months after (T1).
  Interventions: Other: Solid Meal
- Liquid Meal (Other): Participants in this group will be administered only liquid meals on both study visits completed before surgery (T0) and 12-15 months after (T1).
  Interventions: Other: Liquid Meal

INTERVENTIONS:
Other: Liquid Meal
  Arms: Liquid Meal
Other: Solid Meal
  Arms: Solid Meal

SUMMARY:
Analyze the effect of meal pattern (meal number, frequency, and form) on satiety, gut peptides, insulin, and glucose levels in individuals before and 12-15 months after gastric bypass surgery (GBP).

DETAILED DESCRIPTION:
The main goal is to study the effect of meal number, size and texture on metabolism and incretin levels after GBP. Patients will be studied before GBP (T0) and 12-15 months after GBP (T1). At T0 and T1, patients will come for 2 study days for 8 hours: On one study day, a single meal will be served, on the second study day, three small isocaloric meals, with the order of the conditions randomly assigned. The total amount of calories and the overall nutrient composition will be equivalent between conditions. The meals will be either all solid or all liquid. Patients enrolled in the study will be randomly assigned to solid or liquid test meals.

Gastric emptying will be measured by the acetaminophen test.

ELIGIBILITY:
Inclusion Criteria:

* Severely obese patients undergoing gastric bypass surgery (GBP)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2010-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Changes in gut peptides after gastric bypass, during either a liquid or solid meal, or single or multiple isocaloric meals. | 1 month before GBP Surgery, and 12-15 months post surgery
Changes in diet induced thermogenesis after gastric bypass, during either a liquid or solid meal, or single or multiple isocaloric meals. | 1 month before GBP surgery, and 12-15 months post surgery
Changes in insulin levels after gastric bypass, during either a liquid or solid meal, or single or multiple isocaloric meals. | 1 month before GBP surgery, 12-15 months post surgery
Changes in glucose levels after gastric bypass, during either a liquid or solid meal, or single or multiple isocaloric meals. | 1 month before GBP , 12-15 months post GBP
Changes in satiety after gastric bypass, during either a liquid or solid meal, or single or multiple isocaloric meals. | 1 month before GBP, 12-15 months post GBP

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Laferrere, MD, Principal Investigator — New York Obesity Nutrition Research Center
Locations (1):
- St. Lukes- Roosevelt Hospital- New York Obesity Research Center, New York, New York, United States